CLINICAL TRIAL: NCT00544388
Title: Trial to Compare the Efficacy of Levocetirizine and Cetirizine in Reducing Symptoms of Seasonal Allergic Rhinitis in Ragweed Sensitive Subjects Exposed to Pollen Challenge in an Environmental Exposure Unit (EEU).
Brief Title: Efficacy of Levocetirizine and Cetirizine in Reducing Symptoms of Seasonal Allergic Rhinitis in Ragweed Sensitive Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00379
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Levocetirizine dihydrochloride; Xyzal tablet
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levocetirizine dihydrochloride

SUMMARY:
Controlled conditions of the EEU allow a reliable assessment of the efficacy and a determination of the action onset, action intensity and duration of effect of levocetirizine and cetirizine in order to establish the relative efficacy of these two drugs available for the treatment of SAR.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, aged >= 16 years
* seasonal allergic rhinitis that required pharmacologic therapy each year during the last 2 ragweed pollen seasons
* documented seasonal allergy to ragweed pollen
* total symptom score of at least 18 points.

Exclusion Criteria:

* nasal anatomic deformities ? 50% obstruction
* acute sinusitis within 30 days of Period 2
* initiated or advanced an immunotherapy regimen
* immunotherapy injections within 48 hours of pollen exposure
* impaired hepatic function
* history of malignancy
* intolerance to histamines
* asthma requiring medication more than occasionally

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2004-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in major symptom complex score over Period 2 (21-29 hours after drug intake on Day 2).

SECONDARY OUTCOMES:
Mean change from baseline in MSC score over each 2-hour interval.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma